CLINICAL TRIAL: NCT01543815
Title: Well-Being Therapy for Psychological Distress and Enhancing Healthy Behaviors With Personalized Mobile Technology in Cardiac Patients: a Randomized Controlled-trial Study Protocol
Brief Title: Well-Being Therapy by Personalized Mobile Technology Program for Psychological Distress and Promote Healthy Behaviors
Acronym: WELL-ME
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Bergamo (Other)
Responsible Party: Principal Investigator, Angelo Compare, Prof., University of Bergamo
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NCT00289921; 029399 (Other: EU)
Record Dates: First submitted 2012-02-28; First posted 2012-03-05 (Estimated); Last update posted 2012-03-06 (Estimated); Status verified 2011-12

CONDITIONS: Psychological Distress
Keywords: Psychological Distress; Depression; Anxiety; Well-Being Therapy; Heart Failure; Quality of Life; Adherence
MeSH Terms: conditions — Depression; Anxiety Disorders; Heart Failure | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- WBT-WEB (Experimental): Well-Being Therapy based on Web Mobile technology
  Interventions: Behavioral: Well-Being Therapy based on Web Mobile Technology
- CBT (Active Comparator): Cognitive Behavior Therapy
  Interventions: Behavioral: Cognitive Behavior Therapy
- CM (No Intervention): Standardized Care Management
  Interventions: Other: Standardized Care Management

INTERVENTIONS:
Behavioral: Well-Being Therapy based on Web Mobile Technology — The techniques included in WBT may be used in overcoming impairments in environmental mastery, purpose in life, personal growth, autonomy, self-acceptance and positive relations with others.
  Arms: WBT-WEB
Behavioral: Cognitive Behavior Therapy — CBT involves several essential features: identifying and correcting inaccurate thoughts associated with depressed feelings (cognitive restructuring); helping patients to engage more often in enjoyable activities (behavioral activation); enhancing problem-solving skills; providing instruction and guidance in specific strategies for solving problems.
  Arms: CBT
Other: Standardized Care Management — CM will consist of reviewing the patients' clinical status, and providing the patient with support and advice if necessary.
  Arms: CM

SUMMARY:
The WELL-ME study is a three-arm randomized controlled clinical trial (RCT). The aim of this RCT is to compare the effectiveness of the Well Being Web Based Therapy (WBT-Web) with the gold standard CBT (Cognitive Behavior Therapy) and standard clinical procedure of patients' management (CM) for psychological distress and promotion of healthy behaviors in Cardiac Patients.

DETAILED DESCRIPTION:
Cardiac disease (CD) affects millions of European and Americans and new diagnosis rates are expected to almost triple over the next 30 years as our population ages. Affective disorders including clinical depression, anxiety and psychological distress are common in patients with CD. Furthermore, the presence of these disorders significantly impacts quality of life, adherence to medical prescription and healthy behaviors. The prevalence of depression, ranging from 11% to 25% among heart disease outpatients and 35% to 70% among those who are hospitalized. Psychological depression appears to be an important predictor of rehospitalization among persons who have been admitted with coronary artery disease. In addition, depression in patients with heart failure was found to be associated with the course of the disease and its prognosis. The high prevalence of psychological distress among the population of patients with heart failure, along with the broad impact on the patient's quality of life, requires attention to detail and the implementation of interventions aimed at reducing levels of distress. Very few studies describe interventions aimed at alleviating distress in patients with heart failure. Cognitive Behavioral Therapy (CBT) is reported to improve both the functional and emotional levels of these patients, resulting in the relief of their symptoms of depression. Recently Well Being Therapy WBT) have showed promising outcomes findings for depression and distress. There is a need to treat patients in their real life setting. Recent technological innovations in the ICT provide to monitor and treat the patient at a distance outside the hospital. The aim in this study is to study the effectiveness of the WBT-WEB in reducing psychological distress, and improving QoL, healthy behaviors and medical adherence in HR compared to a CBT and standard clinical procedure of patients' management (CM). The same protocol will be carried out in two centres (Hospital de Terrassa, Barcelona, Spain; National and Kapodistrian University of Athens, Greece). 300 patients diagnosed with cardiac disease, and with psychological distress, assessed by Hospital Anxiety and Depression Scale (HADS) will be randomized to one of three treatment groups: 1) WBT-WEB; 2) CBT and 3) CM. A one-year follow-up will be performed. It is expected that WBT-WEB may significantly decrease psychological distress and increase QoL, healthy behaviors and medical adherence at follow-up compared to clinical management.

ELIGIBILITY:
Inclusion Criteria:

* Cardiac Diseases
* a current diagnosis of at least one of the following: major or minor depression, dysthymia, anxiety according, to DSM-IV criteria, and HADS criteria
* Mini-Mental State Examination score higher than 24
* written informed consent provided by the patient to participate

Exclusion Criteria:

* uncertain prognosis for 12 months due to other conditions
* acute coronary disease in recent months.
* existence of another life-threatening illness of the patient (such as active cancer, chronic kidney failure).
* severe neurological problem (Brain syndrome / orientation problem/ difficult peripheral neuropathy).
* severe mental illness (active psychosis / suicide risk / severe dementia).
* linguistic limitations (such as stuttering / untreated audio impairment).
* a significant functional problem (such as unconsciousness / connection to respiration device / confined to a wheelchair or bed / severe walking disability / needs help with complete basic daily activities).
* objective limit that endangers liability for participation in the seven meetings (such as remote residential / tourist / convict / drug addict).

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 400 (Actual)
Dates: Start 2006-01; Primary Completion 2009-02 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Psychological distress | Within one year after the treatment
  Depression, Anxiety, and well-being improvements (Psychological Distress Reduction)

SECONDARY OUTCOMES:
Quality of Life | Within one year after the treatment
  Quality of Life
Medical Adherence | Within one year after the treatment
Promotion of Healthy Lifestyle | Within one year after the treatment
  Promotion of Healthy Lifestyle

CONTACTS AND LOCATIONS:
Overall Officials: Angelo Compare, Ph.D, Principal Investigator — University of Bergamo

REFERENCES:
- [Derived] Compare A, Kouloulias V, Apostolos V, Pena WM, Molinari E, Grossi E, Efstathios E, Carenini M. WELL.ME - Wellbeing therapy based on real-time personalized mobile architecture, vs. cognitive therapy, to reduce psychological distress and promote healthy lifestyle in cardiovascular disease patients: study protocol for a randomized controlled trial. Trials. 2012 Sep 3;13:157. doi: 10.1186/1745-6215-13-157. PMID 22943627 (Retraction: PMID 30572914 Trials. 2018 Dec 20;19(1):692)